CLINICAL TRIAL: NCT00005753
Title: Pharmacological and Behavioral Treatment of Insomnia
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5100; R29HL059387 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-02

CONDITIONS: Lung Diseases; Sleep; Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Lung Diseases; Sleep Initiation and Maintenance Disorders

SUMMARY:
to develop the maximally effective treatment strategy for chronic sleep-onset insomnia and to reduce its impact on psychological functioning, health, and economic sequelae.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The study examined the relative efficacy of a pharmacologic, cognitive behavioral, and conjoint pharmacological/behavioral intervention for chronic sleep-onset insomnia. Sixty-three medication-free, chronic sleep-onset insomniacs completed evaluations, baseline sleep diaries, daytime functioning and mood inventories and home-based objective sleep assessments (OSA). Subjects were then randomized to one of four interventions: 1) six week Zolpidem intervention (D for drug); 2) six week multifactor behavioral intervention (B for behavioral); 3) six week conjoint Zolpidem and multifactor behavioral intervention (DB); and 4) placebo medication intervention (P for placebo). The main outcome measures were sleep-onset latency as measured by sleep diaries; secondary measures included sleep diary measures of sleep efficiency and total sleep time, objective measures of sleep variables (Nightcap sleep monitor recorder), and measures of daytime functioning.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-06; Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Jacobs — Beth Israel Deaconess Medical Center

REFERENCES:
- [Background] Jacobs GD, Pace-Schott EF, Stickgold R, Otto MW. Cognitive behavior therapy and pharmacotherapy for insomnia: a randomized controlled trial and direct comparison. Arch Intern Med. 2004 Sep 27;164(17):1888-96. doi: 10.1001/archinte.164.17.1888. PMID 15451764